CLINICAL TRIAL: NCT00137683
Title: Colorectal Cancer Control in Appalachian Churches
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: West Virginia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-9998; U57/CCU320638
Record Dates: First submitted 2005-08-27; First posted 2005-08-30 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Cancer
Keywords: screening; prevention; community health education
MeSH Terms: conditions — Colorectal Neoplasms; Health Education

INTERVENTIONS:
Behavioral: one-on-one education, group education, small media

SUMMARY:
The purpose of this project is to conduct a community-based intervention and evaluate the independent and combined effects of two intervention strategies on primary and secondary prevention of colorectal cancer (CRC) among members of rural Appalachian churches. The sampling frame consists of all of the churches in a 7 county area of western West Virginia. Eligible churches will have at least 180 active members, will not share a common pastor, and will have no CRC control activities. Using a 2x2 experimental design, churches will be divided into two separate clusters, those with and without an existing parish nurse program. Then churches from each cluster will be randomized to one of two conditions, a natural helper or a control condition.

DETAILED DESCRIPTION:
The purpose of this project is to conduct a community-based intervention and evaluate the independent and combined effects of two intervention strategies on primary and secondary prevention of colorectal cancer (CRC) among members of rural Appalachian churches. Many regions of Appalachia have high poverty, low education, and high unemployment. Health disparities are great in this region and social and behavioral factors put many individuals at high risk for increased mortality from CRC.

The sampling frame consists of all churches in a 7 county area of western West Virginia. Eligible churches will have at least 180 active members, will not share a common pastor, and have no CRC control activities. Using a 2x2 experimental design, churches will be divided into two separate clusters, those with and without an existing parish nurse program. Then churches from each cluster will be randomized to one of two conditions, a natural helper or control condition.

Eligible church members will be adult males and females who are identified through member lists provided by the recruited churches. Because the primary outcome variable is CRC screening, at least half of the recruited church members must be age 50 and older, report no history of CRC, and have not recently completed CRC screening. Interested members will be asked to complete an informed consent form detailing participation in either the intervention or control arm of the study. The control group will be offered other health promotion interventions through the church and the CRC educational materials after data collection is completed.

Data will be collected before and after the intervention activities. Study participants will complete a paper and pencil survey at the church at each measurement point (baseline, follow-up). The baseline survey will assess sociodemographics, psychosocial information, stage of change, self-efficacy, health beliefs, barriers to change, health behavior knowledge and practices involving diet, physical activity, and CRC screening. The follow-up survey will assess body mass index, dietary intake, physical activity level, and CRC screening by FOBT, flexible sigmoidoscopy, and colonoscopy.

The primary hypothesis to be tested is that the combination of these two community-based intervention strategies will be most effective overall. To evaluate the effectiveness of the intervention strategies, the proportions in outcome measures between each intervention, the combined intervention, and control groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Members of church congregations in the Ohio River Valley of West Virginia

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-09; Study Completion 2005-03

PRIMARY OUTCOMES:
colorectal cancer screening

SECONDARY OUTCOMES:
physical activity
diet
knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Irene Tessaro, DrPH, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States